CLINICAL TRIAL: NCT01639144
Title: Use of Platelet-Rich Plasma (PRP) and Platelet-Poor Plasma (PPP) to Prevent Infection and Delayed Wound Healing After Elective Foot and Ankle Surgery in Healthy Adults
Brief Title: Use of Platelet-Rich Plasma (PRP) and Platelet-Poor Plasma (PPP) to Prevent Infection and Delayed Wound Healing
Acronym: PRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gary M. Kiebzak, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Gary M. Kiebzak, Ph.D., Clinical Research Administrator, UHZ Sports Medicine Institute
Organization: UHZ Sports Medicine Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 12-024
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Results first posted 2015-05-22 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Elective Foot and Ankle Surgery.
Keywords: Infection; delayed wound healing; platelet-rich plasma
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Receiving PRP and PPP. (Active Comparator): Administration of PRP and PPP to surgical site.
  Interventions: Biological: PRP and PPP
- Control (No Intervention): Group not receiving autogenous PRP and PPP.

INTERVENTIONS:
Biological: PRP and PPP — Autogenous PRP and PPP
  Arms: Receiving PRP and PPP.

SUMMARY:
The purpose of this study is to see if applying PRP and PPP to surgical sites and the closing incision helps prevent infection and slow wound healing.

DETAILED DESCRIPTION:
This will be a prospective, randomized study with patients blinded to either receiving platelet-rich plasma (PRP) and platelet-poor plasma (PPP) treatment or no treatment. We hypothesize that the antimicrobial properties of PRP and barrier properties of PPP (acting like a tissue sealant) will serve to inhibit deep incisional surgical site infection and help prevent delayed wound healing within 60 days of surgery. Thus, the incidence of infection and delayed wound healing will be lower in patients receiving PRP and PPP compared to patients who do not receive PRP and PPP. However, due to clinical equipoise, we do not know for certain that PRP and PPP is truly effective. The cost of preparing PRP and PPP is substantial, and involves a blood draw that would not otherwise be done. Thus, it is important to know if this treatment is effective or not.

ELIGIBILITY:
Inclusion Criteria:

* Elective foot and ankle surgery.

Exclusion Criteria:

* Younger than 18 years, older than 80 years of age.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2012-07; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary M Kiebzak, Ph.D., Study Director — Center for Research & Grants
Locations (1):
- UHZ Sports Medicine Institute, Coral Gables, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Receiving PRP and PPP. | Control
Started | 260 | 255
Completed | 250 | 250
Not Completed | 10 | 5
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Physician Decision | 2 | 0
Not completed — Met postoperative exclusion criteria | 4 | 3

BASELINE CHARACTERISTICS:
Population: Patients having foot and/or ankle surgery.
Groups:
- Total: Total of all reporting groups
Arm/Group | Receiving PRP and PPP. | Control | Total
Number analyzed (Participants) | 250 | 250 | 500
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 182 | 182 | 364
  >=65 years | 68 | 68 | 136
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 163 | 324
  Male | 89 | 87 | 176
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 250 | 250 | 500
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 250 | 250 | 500
Region of Enrollment [Number; unit: participants]
  United States | 250 | 250 | 500
Diabetes, rheumatoid arthritis, smoking = risk factors for healing [Number; unit: participants]
  Diabetes, rheumatoid arthritis, smoking | 40 | 42 | 82
  No known risk factors for healing | 210 | 208 | 418

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Infection and Delayed Wound Healing.
Description: Postoperative deep incisional surgical site infection and delayed wound healing (lack of primary healing of skin edges typically with wound secretion).
Time Frame: Infection: 30 days after surgery. Delayed wound healing: 60 days.
Population: Patients have foot and/or ankle surgery.
Measure: Number; unit: participants
Arm/Group | Receiving PRP and PPP. | Control
Number analyzed (Participants) | 250 | 250
participants
  Deep surgical site infection | 2 | 1
  Delayed wound healing | 17 | 17

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | Receiving PRP and PPP. | Control
Serious Adverse Events (participants affected / at risk) | 0/250 | 0/250
Other Adverse Events (participants affected / at risk) | 0/250 | 0/250

LIMITATIONS AND CAVEATS:
Originally intended to enroll more patients but due to apparent lack of effect of PRP treatment, enrollment was truncated to n = 250 per study group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes